CLINICAL TRIAL: NCT00964028
Title: Safety and Reactogenicity of GSK Biologicals' DTPa-IPV/Hib (Infanrix™-IPV/Hib) in Infants
Brief Title: Safety Study of GSK Biologicals' DTPa-IPV/Hib (Infanrix™-IPV/Hib)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 112065
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2017-04

CONDITIONS: Haemophilus Influenzae Type b; Acellular Pertussis; Diphtheria; Tetanus; Poliomyelitis
Keywords: Combined vaccine
MeSH Terms: conditions — Haemophilus Infections; Diphtheria; Tetanus; Poliomyelitis

ARMS (2):
- INFANRIX-IPV/HIB M2-M3-M4 GROUP (Experimental): Healthy male or female subjects between and including 60 and 90 days of age at the time of the first vaccination, received 3 doses of Infanrix-IPV/Hib™ vaccine at 2, 3 and 4 months of age (M2-M3-M4), administered intramuscularly into the upper right side of the thigh.
  Interventions: Biological: Infanrix™-IPV/Hib
- INFANRIX-IPV/HIB M3-M4-M5 GROUP (Experimental): Healthy male or female subjects between and including 60 and 90 days of age at the time of the first vaccination, received 3 doses of Infanrix-IPV/Hib™ vaccine at 3, 4 and 5 months of age (M3-M4-M5), administered intramuscularly into the upper right side of the thigh.
  Interventions: Biological: Infanrix™-IPV/Hib

INTERVENTIONS:
Biological: Infanrix™-IPV/Hib — Intramuscular, three doses

SUMMARY:
This study will evaluate the safety and reactogenicity of Infanrix-IPV/Hib given as a three-dose primary vaccination course to healthy infants at 2-3-4 or 3-4-5 months of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female infant between, and including, 60 and 90 days of age at the time of the first study visit.
* Born after a gestation period of 36 to 42 weeks inclusive.
* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* Written informed consent obtained from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs since birth.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Administration of a vaccine not foreseen by the study protocol within 30 days prior to vaccination, or planned administration during the study period, with the exception of hepatitis B vaccine.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Evidence of previous or intercurrent diphtheria, tetanus, pertussis, poliomyelitis and/or Hib disease.
* Previous vaccination against diphtheria, tetanus, pertussis, poliovirus and/or Haemophilus influenzae type b diseases.
* History of seizures or progressive neurological disease.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness.

The following condition is temporary or self-limiting and a subject may be vaccinated once the condition has resolved and no other exclusion criteria are met:

• Current febrile illness or axillary temperature > 37.0 ºC or other moderate to severe illness within 24 hours of study vaccine administration.

Ages: 60 Days to 90 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2009-12-01; Primary Completion 2010-04-12 (Actual); Study Completion 2010-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Wuzhou, Guangxi, China

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following steps occurred: check for inclusion/exclusion criteria, contraindications/precautions, medical history of the subjects and signing informed consent forms.
Groups:
- Infanrix-IPV/Hib M2-M3-M4 Group: Healthy male or female subjects between and including 60 and 90 days of age at the time of the first vaccination, received 3 doses of Infanrix-IPV/Hib vaccine at 2, 3 and 4 months of age (M2-M3-M4), administered intramuscularly into the upper right side of the thigh.
- Infanrix-IPV/Hib M3-M4-M5 Group: Healthy male or female subjects between and including 60 and 90 days of age at the time of the first vaccination, received 3 doses of Infanrix-IPV/Hib vaccine at 3, 4 and 5 months of age (M3-M4-M5), administered intramuscularly into the upper right side of the thigh.
Period: Overall Study
Arm/Group | Infanrix-IPV/Hib M2-M3-M4 Group | Infanrix-IPV/Hib M3-M4-M5 Group
Started | 25 | 25
Completed | 25 | 24
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Infanrix-IPV/Hib M2-M3-M4 Group | Infanrix-IPV/Hib M3-M4-M5 Group | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 10.1 (1.36) | 14.2 (1.18) | 12.15 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 18 | 14 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian heritage | 24 | 25 | 49
  Asian-Japanese heritage | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any local symptom regardless of intensity grade.
Time Frame: During the 4-day (Days 0-3) follow-up period after each dose and across doses
Population: The analysis was performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV/Hib M2-M3-M4 Group | Infanrix-IPV/Hib M3-M4-M5 Group
Number analyzed (Participants) | 25 | 25
Participants
  Any Pain, Dose 1 | 4 | 2
  Any Redness, Dose 1 | 2 | 0
  Any Swelling, Dose 1 | 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 25 | 24
  Any Pain, Dose 2 | 1 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 25 | 24
  Any Redness, Dose 2 | 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 25 | 24
  Any Swelling, Dose 2 | 1 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 25 | 24
  Any Pain, Dose 3 | 2 | 1
  Any Redness, Dose 3: number analyzed (Participants) | 25 | 24
  Any Redness, Dose 3 | 2 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 25 | 24
  Any Swelling, Dose 3 | 0 | 0
  Any Pain, Across doses | 4 | 3
  Any Redness, Across doses | 4 | 0
  Any Swelling, Across doses | 2 | 0

2. Primary Outcome: Number of Subjects With Any Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, irritability, loss of appetite and fever [defined as axillary temperature equal to or above 37.0 degrees Celsius (°C)]. Any = occurrence of any general symptom regardless of intensity grade or relationship to vaccination.
Time Frame: During the 4-day (Days 0-3) follow-up period after each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV/Hib M2-M3-M4 Group | Infanrix-IPV/Hib M3-M4-M5 Group
Number analyzed (Participants) | 25 | 25
Participants
  Any Drowsiness, Dose 1 | 9 | 1
  Any Irritability, Dose 1 | 9 | 5
  Any Loss of appetite, Dose 1 | 7 | 1
  Any Fever, Dose 1 | 8 | 8
  Any Drowsiness, Dose 2: number analyzed (Participants) | 25 | 24
  Any Drowsiness, Dose 2 | 3 | 5
  Any Irritability, Dose 2: number analyzed (Participants) | 25 | 24
  Any Irritability, Dose 2 | 6 | 3
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 25 | 24
  Any Loss of appetite, Dose 2 | 3 | 3
  Any Fever, Dose 2: number analyzed (Participants) | 25 | 24
  Any Fever, Dose 2 | 5 | 5
  Any Drowsiness, Dose 3: number analyzed (Participants) | 25 | 24
  Any Drowsiness, Dose 3 | 2 | 0
  Any Irritability, Dose 3: number analyzed (Participants) | 25 | 24
  Any Irritability, Dose 3 | 5 | 4
  Any Loss of appetite, Dose 3: number analyzed (Participants) | 25 | 24
  Any Loss of appetite, Dose 3 | 3 | 1
  Any Fever, Dose 3: number analyzed (Participants) | 25 | 24
  Any Fever, Dose 3 | 7 | 3
  Any Drowsiness, Across doses | 12 | 5
  Any Irritability, Across doses | 15 | 8
  Any Loss of appetite, Across doses | 9 | 4
  Any Fever, Across doses | 13 | 12

3. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 31-day (Days 0-30) follow-up period after each vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV/Hib M2-M3-M4 Group | Infanrix-IPV/Hib M3-M4-M5 Group
Number analyzed (Participants) | 25 | 25
Participants | 16 | 1

4. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the whole study period (from Day 0 until Month 3 or Month 4)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Infanrix-IPV/Hib M2-M3-M4 Group | Infanrix-IPV/Hib M3-M4-M5 Group
Number analyzed (Participants) | 25 | 25
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: during the 31-day (Days 0-30) post-vaccination period. SAEs: during the entire study period (from Day 0 until Month 3/4).
Arm/Group | Infanrix-IPV/Hib M2-M3-M4 Group | Infanrix-IPV/Hib M3-M4-M5 Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 23/25 | 16/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Infanrix-IPV/Hib M2-M3-M4 Group (N=25) | Infanrix-IPV/Hib M3-M4-M5 Group (N=25)
Pyrexia (General disorders) | 5 | 0
Pain (General disorders) | 4 | 3
Redness (General disorders) | 4 | 0
Swelling (General disorders) | 2 | 0
Drowsiness (General disorders) | 12 | 5
Irritability (General disorders) | 15 | 8
Loss of appetite (General disorders) | 9 | 4
Fever (General disorders) | 13 | 12
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 10 | 1
Nasopharyngitis (Infections and infestations) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.